CLINICAL TRIAL: NCT04455061
Title: Intestinal Flora Research Plan for Critically Ill Patients-- Study on the Relationship Between Microbial Disorder and Disease Severity, Prognosis
Brief Title: Intestinal Flora Research Plan for Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-01-01
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-01

CONDITIONS: Gut Microbiota, PICS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
More and more critically ill patients have improved early survival, they have been suffering from organ damage and inflammation for a long time, which is called chronic critical illness (CCI). Among CCI, persistent inflammatory response-immunosuppression-catabolic syndrome (PICS) is a special type of chronic severe disease, and immune paralysis is its main feature. The clinical manifestations are repeated nosocomial infections, malnutrition, muscle loss, and difficulty in wound healing and require long-term emergency medical support, which ultimately leads to patients Repeated nosocomial infections, prolonged hospitalization, and increased mortality.

The gut provides the microbiome with habitat and the nutrients it needs, down-regulates the immune response to form immune tolerance, and promotes its colonization in the intestine.Under physiological conditions, the mutually beneficial symbiosis of the intestine and microorganisms promotes the body's homeostasis. The composition and biodiversity of the microbial community are highly susceptible to various factors, including diet, environment, drugs, infections, inflammation, etc. Especially for acute stress, severe stress, the use of broad-spectrum antibiotics, vasoconstrictors and opioids, intestinal ischemia/reperfusion injury, epithelial cell apoptosis, barrier integrity destruction, gastrointestinal Changes in the motility of the tract, lack of nutrients in the intestinal cavity, etc. All those can lead to rapid changes in the intestinal flora, and this change can last for a long time; manifested by the loss of the richness and diversity of the intestinal microflora (especially the symbiotic flora), The ratio of Bacteroidetes/thickwalled bacteria is severely unbalanced, and a single flora (often a potential pathogen) overgrows, that is, bacterial flora imbalance or microecological disturbance.

At present, for critically ill patients, there are few relevant studies, and currently limited to small-scale, single cross-sectional studies. These studies have uncovered the changes and impacts of intestinal microbiota in critically ill patients in ICU, but they are still in the stage of touching the image of blind people. The relevant mechanisms and dynamic changes and their significance are unclear, requiring large-scale, dynamic, continuous and comprehensive In order to accurately grasp the role of intestinal flora in the development and prognosis of the disease, we hope to accurately control the intestinal flora and achieve effective treatment.

DETAILED DESCRIPTION:
With the improvement and development of medical technology and concepts, the types, progression, and outcomes of critically ill patients have changed dramatically. More and more critically ill patients can successfully escape from the early critical state, and the outbreak of multiple organ failure has been alleviated. However, due to the residual organ dysfunction, the number of cases staying in the intensive care department for a long time is increasing. Both severe trauma and sepsis undergo similar transformations. Although these patients have improved early survival, they have been suffering from organ damage and inflammation for a long time, which is called chronic critical illness (CCI). The definition of CCI includes the number of days of ICU hospitalization greater than or equal to 14 days, evidence of persistent organ dysfunction, and can be measured using components of the 14-day Sequential Organ Failure Assessment (SOFA) score. Even nearly 40% of sepsis patients will develop CCI. These critical survivors continue to recover and support treatment even after being discharged from the hospital, often failing to recover and eventually die. Among them, persistent inflammatory response-immunosuppression-catabolic syndrome (PICS) is a special type of chronic severe disease, and immune paralysis is its main feature. These patients also face several challenges such as persistent inflammatory response, acquired immunosuppression, and high catabolism. The clinical manifestations are repeated nosocomial infections, malnutrition, muscle loss, and difficulty in wound healing and require long-term emergency medical support, which ultimately leads to patients Repeated nosocomial infections, prolonged hospitalization, and increased mortality.

Due to the decline in organ function reserve of elderly patients, chronic diseases of basic heart, lung, kidney and other systems are often combined. After suffering trauma and severe infection, organ function disorders or failures are prone to occur and stay in the ICU ward. With the advent of an aging population, such patients are increasing year by year. It is a heavy burden on society and a huge challenge for the future development and progress of ICU.

The gut flora is involved in a wide range of functions, food digestion, hormone production, and the development and maturation of the immune system. After more than a billion years of co-evolution, a stable symbiotic relationship has been formed between mammals including humans and the gut microbiota. The gut provides the microbiome with habitat and the nutrients it needs, down-regulates the immune response to form immune tolerance, and promotes its colonization in the intestine; accordingly, the gut symbiotic microbiota promotes the health of the body in various ways to form symbiosis Mode: (1) Inhibiting the colonization of pathogenic bacteria by competing for niche and nutrients, producing virulence factors, and secreting bacteriocins, preventing their overgrowth, and protecting the body from pathogen infection, called colonization resistance; (2 ) Promote the proliferation of epithelial cells, secrete antimicrobial peptides and mucus to maintain the integrity of the intestinal barrier; (3) Indirectly regulate the differentiation of innate and adaptive immune cells located in the intestinal epithelial barrier and the whole body, promote the development and maturation of the immune system, and strengthen immune cells Function; (4) Induce extravascular tissue factor-protease activated receptor 1 (TF-PAR1) signal transduction, promote small intestine angiogenesis; (5) participate in hormone signal transduction, regulate intestinal endocrine function; (6) participate in intestinal origin Serotonin (5-HT) metabolism and intestinal neuro-immune cooperation, regulate gastrointestinal motility; (7) produce short-chain fatty acids (SCFAs) by fermenting dietary fiber, improve glucose homeostasis and insulin sensitivity, participate in anti-inflammatory, Promote intestinal motility; (8) Synthesize essential vitamins and neurotransmitters and metabolize bile salts; (9) Participate in body drug metabolism and poison removal. This shows that under physiological conditions, the mutually beneficial symbiosis of the intestine and microorganisms promotes the body's homeostasis. The composition and biodiversity of the microbial community are highly susceptible to various factors, including diet, environment, drugs, infections, inflammation, etc. Especially for acute stress, severe stress, the use of broad-spectrum antibiotics, vasoconstrictors and opioids, intestinal ischemia/reperfusion injury, epithelial cell apoptosis, barrier integrity destruction, gastrointestinal Changes in the motility of the tract, lack of nutrients in the intestinal cavity, etc. lead to rapid changes in the intestinal flora, and this change can last for a long time; manifested by the loss of the richness and diversity of the intestinal microflora (especially the symbiotic flora), The ratio of Bacteroidetes/thickwalled bacteria is severely unbalanced, and a single flora (often a potential pathogen) overgrows, that is, bacterial flora imbalance or microecological disturbance.

The local immune inflammatory storm in the intestine is an important cause of the imbalance of the systemic immune inflammatory response, and the hypothalamic metabolism center is an important target for regulating the body's continuous catabolism. In PICS, immunosuppression, inflammation, and catabolism are mutually causal, forming a vicious circle. So what is the reason for severe patients with different primary diseases to have the same PICS after the acute phase? Are there common pathological changes induced by PICS in severe patients? If further studies can be made to clarify the initiating factors of PICS and the path of occurrence and development of PICS, it is undoubtedly a new breakthrough in the treatment of PICS and the "fundamental" way to reduce the mortality of PICS patients. Combining our previous research results, applicants speculate as follows:

1. The intestinal tract is the "promoting point" for the occurrence of PICS in severely ill patients, and it is also the "central organ" that promotes the development of the disease; 2. The disturbance of the micro-ecology of the intestinal tract is an important reason for causing PICS in the body (and may even be the decisive factor) ; 3. Correction of intestinal microecological disturbances can effectively block the path of PICS development.

For the above ideas, specific explanations are as follows:

1. The intestine may be the "promoting point" for PICS in critically ill patients, and it is also the "central organ" that promotes the development of the disease. The reasons are as follows:

   * Our previous studies showed that acute gastrointestinal dysfunction is common in severe patients. Whether it is local simple abdominal exposure injury or systemic ischemia-reperfusion injury, it can cause acute gastrointestinal dysfunction; ②The intestine is not only the main organ of digestion and absorption, but also the body's largest immune organ (adult). When the intestine is acutely damaged, the intestine can affect the nutritional metabolism center of the hypothalamus through Grelin and other hormones, leading to refractory catabolism and exogenous nutrition. At the same time, the local inflammatory reaction of the intestinal tract can also cause an imbalance of the body's immune inflammatory response. In addition, changes in central metabolism in critically ill patients are related to hypothalamic inflammation (indicating that the intestine is "capable" to become the central organ that promotes the occurrence and development of PICS).

Intestinal microecological disturbance is an important cause of PICS Under normal physiological conditions, the intestine has powerful barrier functions, such as physical barrier, chemical barrier, immune barrier, and biological barrier. Especially its biological barrier function plays an important role in the body's metabolism and immunity. There is a stable symbiotic relationship between the human body and the intestinal microbiota. The intestine provides the microbiome with habitat and the nutrients it needs to downregulate the immune response to form immune tolerance and promote its colonization in the intestine; accordingly, the physiological state Next, the gut symbiotic microbiota also maintains the body's health in various ways [2]. The intestine and microorganisms are symbiotic and promote the body's homeostasis. However, the composition and biodiversity of the microbial community are highly susceptible to various factors, including diet, environment, drugs, infections, inflammation, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Expect to stay in the ICU for more than 7 days after enrollment;
3. Initial disease, not receiving ICU special treatment;

Exclusion Criteria:

1. Does not meet the inclusion criteria;
2. Complicated with perianal infection, intestinal fistula, short bowel syndrome, chronic severe gastrointestinal disease;
3. Patients with malignant tumors undergoing chemotherapy and radiotherapy;
4. Taking probiotic preparations within the past 3 months, etc. Intestinal flora regulator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to further understand and grasp the relationship between the intestinal microflora in critically ill patients, the relationship with the progression of critical illness, the outcome of the disease and the final prognosis, it is now planned to analyze the dynamic intestinal microflora changes in critically ill patients through 16SrRNA technology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | up to 28 days after hospitalized.
  The patient's 28-day mortality rate is the survival rate from the onset to the disease at 28 days, compared with the total number of illnesses, to assess the severity of the disease

SECONDARY OUTCOMES:
the duration of intensive care unit | Up to 8 weeks
  time for patients treatment in intensive care unit is patient total treated days in intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Chen X, Li H, Huang S, Chen M, Huang S, Zhu Z, You Y, Xu G, Wang Y, Wang R, Yu W. ROLE OF CHANGES IN LIPOPROTEINS, LIPIDOMES, AND GUT MICROBIOTA IN THE PATHOGENESIS OF PERSISTENT INFLAMMATION, IMMUNOSUPPRESSION, AND CATABOLISM SYNDROME: A PROSPECTIVE COHORT STUDY. Shock. 2025 Sep 1;64(3):322-331. doi: 10.1097/SHK.0000000000002634. PMID 40844181